CLINICAL TRIAL: NCT05903690
Title: Safety and Tolerance of RAG-17 in Amyotrophic Lateral Sclerosis Patients With SOD1 Gene Mutation
Acronym: CREATION
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Ractigen Therapeutics. (Other)
Responsible Party: Principal Investigator, yilong Wang, Vice-President of Beijing Tiantan Hospital,Chief Scientist of Neurology Center, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX-A-2023004
Record Dates: First submitted 2023-05-07; First posted 2023-06-15 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Gene Mutation
Keywords: RAG-17; SOD1 Gene Mutation; Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RAG-17 (Experimental): Doses of RAG-17 will range from a minimum of 60 mg to the maximum tolerated dose (MTD). Dosing once every two weeks, starting from 60 mg, with dose escalation. After reaching the tolerated dose, a fixed dose of the drug is given once every two months for continuous treatment, and the total treatment cycle is 8 months.
  Interventions: Drug: RAG-17

INTERVENTIONS:
Drug: RAG-17 — RAG-17 60mg is used

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability and pharmacokinetics of RAG-17 in adult amyotrophic lateral sclerosis (ALS) patients with SOD1 mutation. Patients will receive drug treamtent via dose escalation which ranging from minimum of 60 mg to the maximum tolerated dose (MTD), after reaching the tolerated dose, a fixed dose of the drug is given once every two months for continuous treatment, and the total treatment cycle is 8 months. The duration of this study is two years.

DETAILED DESCRIPTION:
This study is an open-label, single center, first-in-Human dose escalation study to evaluate the safety, tolerability and pharmacokinetics of RAG-17 in adultamyotrophic lateral sclerosis (ALS) patients with SOD1 mutation via dose escalations. Patients will receive 60mg of RAG-17 firstly, within 14 days after the first administration, the subject has no adverse event (AE) and serious adverse event (SAE), the subject can accept dose escalation every 30mg/14 days of observation period. 3 to 4 dose escalations are planned to reach the dose limiting toxicity (DLT), with optimal doses for continual 6-month treatment cycles. For the dose of subsequent continuous treatment, an optimal dose between the safe dose and the maximum tolerated dose (MTD) is selected as the continuous treatment dose. SAS software is used for safety analysis. The sample size of this study is 6 ALS patients with SOD1 mutation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are judged by professional medical staff to still be able to carry out the clinical trial project cycle;
* 18 years old ≤ age ≤ 75 years old, males or females;
* ALS patients with confirmed SOD1 gene mutations document (known SOD1 mutation sites and related disease progression have been reported);
* Forced vital capacity ≥ 50% of predicted vital capacity during the screening period;
* Diagnosis of confirmed or probable familial or sporadic ALS in accordance with the revised EI Escorial diagnostic criteria for amyotrophic lateral sclerosis of the World Federation of Neurology;
* The patient or patient's legal representative clearly understands and voluntarily participates in the study and signs the informed consent form;
* Subjects (including male subjects) are willing to have no birth plan and voluntarily take effective contraceptive measures during the entire study period and within 3 months after the end of the study, and have no plan to donate sperm or eggs.

Exclusion Criteria:

* Patients with SOD1 mutations occurring at nucleotides 44 to 66 (calculated from the start of SOD1 protein translation), patients with P.F21C mutation;
* Patients who have previously received or are currently receiving Tofersen treatment;
* HIV test positive or history of positive tests;
* Positive hepatitis C virus antibody or history of positive tests;
* Active hepatitis B infection (positive hepatitis B surface antigen and/or positive hepatitis B core antibody);
* Have used other investigational drugs within 1 month or within 5 drug half-lives;
* Diseases and deformities of the lumbar spine;
* Have other conditions known to be associated with motor neuron dysfunction that may confuse or obscure an ALS diagnosis;
* Other psychiatric disorders diagnosed according to DSM-V diagnostic criteria, or significant suicide intent;
* With severe hepatic insufficiency, renal insufficiency or severe cardiac insufficiency (severe hepatic insufficiency refers to ALT value≥2.0 times the upper limit of normal value or AST value≥2.0 times the upper limit of normal value; severe renal insufficiency refers to CRE≥1.5 times the upper limit of normal value or eGFR<40mL/min/1.73m2; severe cardiac insufficiency refers to NYHA class 3-4);
* Permanently dependent on ventilator-assisted ventilation;
* History of alcohol and drug abuse;
* Patients who are pregnant, breast-feeding, or who are likely to become pregnant and plan to become pregnant;
* Patients participating in other clinical trials or using other biological agents, drugs or devices under investigation;
* Patients who have received any vaccinations within 28 days;
* Contraindications to MRI (eg, claustrophobia);
* Unable to be cooperative and complete the follow-up due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Adverse events (AE) and serious adverse events (SAE) | Within 240 days after treatment
  The incidence of adverse events (AE) and serious adverse events (SAE) within 240 days after the first injection of RAG-17, and number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) V5.0
Clinical laboratory examination index | Before RAG-17 treatment and within 240 days after treatment
  Monitor the abnormal change of clinical laboratory Index generated from general examination results before RAG-17 treatment, and within 240 days after the first injection of RAG-17, which including blood testing and urine testing. Eventually to determine the safety and tolerability of RAG-17 on adult ALS patients.
Physiological Parameter-Vital Sign: Body Temperature | Within 240 days after treatment
  Change in vital signs are monitored within 240 days after RAG-17 treatment to determine the safety and tolerability of RAG-17 on adult ALS patients. Vital sign that is measured including body temperature in degree Celsius.
Physiological Parameter-Vital Sign: Pulse Rate | Within 240 days after treatment
  Change in vital signs are monitored within 240 days after RAG-17 treatment to determine the safety and tolerability of RAG-17 on adult ALS patients. Vital sign that is measured including pulse rate in beats per minute.
Physiological Parameter-Vital Sign: Respiration Rate | Within 240 days after treatment
  Change in vital signs are monitored within 240 days after RAG-17 treatment to determine the safety and tolerability of RAG-17 on adult ALS patients. Vital sign that is measured including respiration rate in breaths per minute.
Physiological Parameter-Vital Sign: Blood Pressure | Within 240 days after treatment
  Change in vital signs are monitored within 240 days after RAG-17 treatment to determine the safety and tolerability of RAG-17 on adult ALS patients. Vital sign that is measured including blood pressure in mmHg.
Physiological Parameter-Vital Signs: Height, Hip Circumference and Waist | Within 240 days after treatment
  Change in vital signs are monitored within 240 days after RAG-17 treatment to determine the safety and tolerability of RAG-17 on adult ALS patients. Vital signs that are measured including height, hip circumference and waist in centimeter.
Physiological Parameter-Vital Signs: Weight | Within 240 days after treatment
  Change in vital signs are monitored within 240 days after RAG-17 treatment to determine the safety and tolerability of RAG-17 on adult ALS patients. Vital sign that is measured including body weight in kilogram.
Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R) | Within 240 days after treatment
  Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R) is a questionnaire-based scale that is used to measure the change in functional impairment of adult ALS patients within 240 days after RAG-17 treatment. ALSFRS-R scale measures 12 aspects of physical function, and each function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0.
Neurological examinations | Within 240 days after treatment
  Incidence rate of abnormalities in neurological examinations within 240 days after RAG-17 treatment
Heart circulatory system examinations | Within 240 days after treatment
  Incidence rate of abnormalities in heart circulatory system examinations within 240 days after RAG-17 treatment
Respiratory system examinations | Within 240 days after treatment
  Incidence rate of abnormalities in respiratory system examinations within 240 days after RAG-17 treatment
Abdominal examinations | Within 240 days after treatment
  Incidence rate of abnormalities in abdominal examinations within 240 days after RAG-17 treatment
ECG results | Within 240 days after treatment
  Incidence rate of abnormalities in ECG results within 240 days after RAG-17 treatment

SECONDARY OUTCOMES:
SOD1 protein levels | baseline, day 15, day 29, day 60, day 120, day 180 and day 240
  Changes of SOD1 protein levels in cerebrospinal fluid from baseline on day 15, day 29, day 60, day 120, day 180 and day 240 of adult ALS patients after RAG-17 treatment
Plasma neurofilament light (NFL) levels | baseline, day 1, day 15, day 29, day 60, day 120, day 180 and day 240
  Changes in plasma neurofilament light (NFL) levels from baseline on day 1, day 15, day 29, day 60, day 120, day 180 and day 240 in adult ALS patients after RAG-17 treatment
Pharmacokinetic Changes of RAG-17 | day 1, day 15, day 29, day 60, day 120, day 180 and day 240
  Pharmacokinetic Parameter changes of RAG-17 in Plasma: Maximum Observed Concentration (Cmax) on day1, day15, day29, day60, day120, day180 and day240 in adult ALS patients after RAG-17 treatment
Pharmacokinetic Changes of RAG-17 | day 1, day 15, day 29, day 60, day 120, day 180 and day 240
  Pharmacokinetic Parameter changes of RAG-17 in Plasma: Time to Reach Maximum Observed Concentration (Tmax) on day1, day15, day29, day60, day120, day180 and day240 in adult ALS patients after RAG-17 treatment
Pharmacokinetic Changes of RAG-17 | day 1, day 15, day 29, day 60, day 120, day 180 and day 240
  Pharmacokinetic Parameter changes of RAG-17 in Plasma: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) on day1, day15, day29, day60, day120, day180 and day240 in adult ALS patients after RAG-17 treatment
Pharmacokinetic Changes of RAG-17 | day 1, day 15, day 29, day 60, day 120, day 180 and day 240
  Pharmacokinetic Parameter changes of RAG-17 in Plasma: Area Under the Concentration-time Curve From Time Zero to the Time of the Last Measurable Concentration (AUClast) on day1, day15, day29, day60, day120, day180 and day240 in adult ALS patients after RAG-17 treatment
Pharmacokinetic Changes of RAG-17 | day 1, day 15, day 29, day 60, day 120, day 180 and day 240
  Pharmacokinetic Parameter changes of RAG-17 in Plasma: Apparent Terminal Elimination Half-life (t1/2) on day1, day15, day29, day60, day120, day180 and day240 in adult ALS patients after RAG-17 treatment
Mechanical ventilation | From day1 to day240
  Time to invasive mechanical ventilation in adult ALS patients treated with RAG-17
Death | From randomization date to date of death from any cause. The assessment period is up to 8 months
  Time of death in adult ALS patients treated with RAG-17

OTHER OUTCOMES:
Lung function (including forced vital capacity) | day 15, day 29, day 90, day 180, and day 240
  Changes in lung function (including forced vital capacity) in adult ALS patients treated with RAG-17 on day 15, day 29, day 90, day 180, and day 240
Severity of Fatigue (Fatigue Severity Scale - FSS) | day 15, day 29, day 90, day 180, and day 240
  Fatigue Severity Scale(FSS) is a questionnaire-based scale that is used to measure the change in severity of fatigue in adult ALS patients on day 15, day 29, day 90, day 180, and day 240 after RAG-17 treatment. FSS scale is 9-items questionnaire, and each item is scored on a 7 points scale from 1 (strongly disagree) to 7 (strongly agree). The minimum score in total is 9 points, and the maximum score possible is 63. The higher the score means the greater fatigue severity.
Muscle strength (Medical Research Council Scale - MRC Scale) | day 15, day 29, day 90, day 180, and day 240
  Medical Research Council Scale (MRC Scale) is an assessment that is used to measure the change in muscle strength of abductor pollicis brevis muscle, abductor digiti minimi, and tibial anterior muscle in adult ALS patients treated with RAG-17 on day 15, day 29, day 90, day 180, and day 240. MRC Scales ranges from grade 0 to grade 5, where grade 0 means no muscle contraction, grade 5 means muscle has full strength.
Electromyography (EMG) measures | day 29, day 90, day 180, and day 240
  Electromyography(EMG) is used to determine the functional performance of muscle and the index change including compound muscle action potential（CAMP）of EMG in adult ALS patients from baseline on day 29, day 90, day 180, and day 240 after RAG-17 treatment
Electromyography (EMG) Measures | day 29, day 90, day 180, and day 240
  Changes in EMG measures (motor unit number index) from baseline on day 29, day 90, day 180, and day 240 after RAG-17 treatment in adult ALS patients
Electromyography (EMG) Measures | day 29, day 90, day 180, and day 240
  Changes in EMG measures (motor unit size index) from baseline on day 29, day 90, day 180, and day 240 after RAG-17 treatment in adult ALS patients
7T magnetic resonance imaging measures | day 29, day 90, day 180, and day 240
  7T magnetic resonance imaging (7T MRI) is used to measure the change in the value of body indexes in adult ALS patients treated with RAG-17 on day 29, day 90, day 180, and day 240.
Kinetic Gait Analysis-Gait Function | day15, day 29, day 90, day 180, and day 240
  Kinetic gait analysis is used to determine the forces created by and during movement, and measurements are collected to further determine the change in gait functions of of adult ALS patients on day 15, day 29, day 90, day 180, and day 240 after RAG-17 treatment.
Kinematic Gait Analysis-Gait Function | day15, day 29, day 90, day 180, and day 240
  Kinematic gait is studied via 3D motion analysis, Construction of the coordinates and orientation of the rigid body segments allow calculation of joint angles of the proximal and distal segment, joint angular velocity, and joint acceleration. Measurements are collected for each joint in all three cardinal planes of motion, and it further measures the change in gait functions of of adult ALS patients on day 15, day 29, day 90, day 180, and day 240 after RAG-17 treatment.
Short Physical Performance Battery (SPPB) - Gait Function | day 15, day 29, day 90, day 180, and day 240
  Short Physical Performance Battery (SPPB) is an objective assessment that is used to measure the change in gait functions including balance, lower extremity strength, and functional capacity of of adult ALS patients on day 15, day 29, day 90, day 180, and day 240 after RAG-17 treatment. The test includes three different assessments: walking, sit-to-stand and balance. A 0- to 12-point scale is used to score the sum of the three assessments with higher point values corresponding with greater levels of physical function and lower disability, and vise versa.
Scale for the Assessment and Rating of Ataxia (SARA) - First Item: Gait | day 15, day 29, day 90, day 180, and day 240
  Scale for the Assessment and Rating of Ataxia (SARA) is a performance based scale that has eight categories to assess different impairments. The first category - gait of SARA is used to measure the change in gait function of adult ALS patients on day 15, day 29, day 90, day 180, and day 240 after RAG-17 treatment. Gait function is scored from 0point (normal) to 8points (unable to walk).
6-meter Walking Test - Gait function | day 15, day 29, day 90, day 180, and day 240
  6-meter walking test is a performance test to assess walking speed over a short distance, which determine the changes in gait function of adult ALS patients on day 15, day 29, day 90, day 180, and day 240 after RAG-17 treatment. The test will be perform in 4 trials, as the first trial is practise trial, and the average of last three trials are calculated.
The Modified Norris Test Score - Functional ability | day 15, day 29, day 90, day 180, and day 240
  The Modified Norris Test Score is a rating scale that is used to measure the change in functional ability of adult ALS patients on day 15, day 29, day 90, day 180, and day 240 after RAG-17 treatment. This scale is composed with two parts: the Limb Norris Scale (21 items) and the Norris Bulbar Scale (13 items), each item is scored from 0 point (cannot do anything) to 3 points (normal).
Amyotrophic Lateral Sclerosis Assessment Questionnaire -40 (ALSAQ-40) - The Quality of Life | day 15, day 29, day 90, day 180, and day 240
  Amyotrophic Lateral Sclerosis Assessment Questionnaire -40 (ALSAQ-40) is a patient self-report health status PRO that is used to measure the changes in the quality of life of adult ALS patients treated with RAG-17 on day 15, day 29, day 90, day 180, and day 240. There are 40 items in ALSAQ-40 with 5 domains: physical mobility (10 items), activities of daily living and independence (10 items), eating and drinking (3 items), communication (7 items), emotional reactions (10 items), each domain has a total score of 100 points, where 0 point means the worst health condition, and 100points means the best health condition.
The EuroQol 5 Dimension 5 Level (EQ-5D-5L)- The Quality of Life | day 15, day 29, day 90, day 180, and day 240
  The EuroQol 5 Dimension 5 Level (EQ-5D-5L) is a self-report survey that is used to measure the changes in the quality of life of adult ALS patients treated with RAG-17 on day 15, day 29, day 90, day 180, and day 240. EQ-5D-5L contains 5 domains including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and each domain is scored on a 5-level severity from Level1(no difficulty) to Level5 (extreme difficulty).
Hamilton Anxiety Scale (HAM-A) - The Quality of Life | day 15, day 29, day 90, day 180, and day 240
  Hamilton Anxiety Scale (HAM-A) is a rating scale that is used to measure the changes in severity of anxiety of adult ALS patients treated with RAG-17 on day 15, day 29, day 90, day 180, and day 240. The scale is composed of 14 items, Each item is scored on a scale of 0 (no symptom) to 4 (severe), with a total score range of 0 to 56, where <7 means no symptom of anxiety, over 24 means mild to moderate severity, >29 means extreme severity.
Hamilton Depression Scale (HAM-D)-The Quality of Life | day 15, day 29, day 90, day 180, and day 240
  Hamilton Depression Scale (HAM-D) is a rating scale that is used to measure the changes in severity of depression of adult ALS patients treated with RAG-17 on day 15, day 29, day 90, day 180, and day 240. For the 17-item version, scores can range from 0 to 54. Scores between 0 and 6 indicate a normal person , scores between 7 and 17 indicate mild depression, scores between 18 and 24 indicate moderate depression, and scores over 24 indicate severe depression.
London ALS Stage - Clinical staging of patients | day 15, day 29, day 90, day 180, and day 240
  London ALS Stage is used to measure the change in clinical stages of adult ALS patients on day 15, day 29, day 90, day 180, and day 240 after RAG-17 treatment. The King's staging system consists of five disease stages, with Stage 5 being death. Stage 4 is nutritional failure.Stages 1-3 are based upon the number of El Escorial central nervous system (CNS) regions involved in the disease, measured by weakness, wasting, spasticity, dysphagia, or dysarthria.
The Milano-Torino (MiToS) Staging - Clinical staging of patients | day 15, day 29, day 90, day 180, and day 240
  The Milano-Torino (MiToS) Staging is used to measure the change in clinical stages of adult ALS patients on day 15, day 29, day 90, day 180, and day 240 after RAG-17 treatment. The Milano-Torino (MiToS) Staging is composed with six stages, where stage 0 is no functional impairment, stage 1 is loss of one type of function, stage 2 is loss of two type of function, stage 3 is loss of three type of function, stage 4 is loss of four type of function, and stage 5 is death.

CONTACTS AND LOCATIONS:
Overall Officials: YiLong Wang, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feldman EL, Goutman SA, Petri S, Mazzini L, Savelieff MG, Shaw PJ, Sobue G. Amyotrophic lateral sclerosis. Lancet. 2022 Oct 15;400(10360):1363-1380. doi: 10.1016/S0140-6736(22)01272-7. Epub 2022 Sep 15. PMID 36116464
- [Background] Chen L, Zhang B, Chen R, Tang L, Liu R, Yang Y, Yang Y, Liu X, Ye S, Zhan S, Fan D. Natural history and clinical features of sporadic amyotrophic lateral sclerosis in China. J Neurol Neurosurg Psychiatry. 2015 Oct;86(10):1075-81. doi: 10.1136/jnnp-2015-310471. Epub 2015 Jun 29. PMID 26124198
- [Background] Rosenbohm A, Liu M, Nagel G, Peter RS, Cui B, Li X, Kassubek J, Rothenbacher D, Lule D, Cui L, Ludolph AC; ALS Registry Swabia Study Group. Phenotypic differences of amyotrophic lateral sclerosis (ALS) in China and Germany. J Neurol. 2018 Apr;265(4):774-782. doi: 10.1007/s00415-018-8735-9. Epub 2018 Feb 1. PMID 29392461
- [Background] Amyotrophic Lateral Sclerosis (ALS) Fact Sheet. National Institute of Neurological Disorders and Stroke. https://www.ninds.nih.gov/amyotrophic-lateral-sclerosis-als-fact-sheet#treatment. October 2022.
- [Background] Miller RG, Jackson CE, Kasarskis EJ, England JD, Forshew D, Johnston W, Kalra S, Katz JS, Mitsumoto H, Rosenfeld J, Shoesmith C, Strong MJ, Woolley SC; Quality Standards Subcommittee of the American Academy of Neurology. Practice parameter update: the care of the patient with amyotrophic lateral sclerosis: drug, nutritional, and respiratory therapies (an evidence-based review): report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2009 Oct 13;73(15):1218-26. doi: 10.1212/WNL.0b013e3181bc0141. PMID 19822872
- [Background] Barrington CJ, Burruano M, Carney C, Choi J, Januska J, Lachuk L, Oskarsson B, Rodriguez C, Speicher L, Tereso G. Addressing the role of edaravone in the management of amyotrophic lateral sclerosis and gaps in care and access: expert panel recommendations. Am J Manag Care. 2021 Aug;27(12 Suppl):S231-S237. doi: 10.37765/ajmc.2021.88732. PMID 34382759
- [Background] Emery AE, Holloway S. Familial motor neuron diseases. Adv Neurol. 1982;36:139-47. No abstract available. PMID 7180680
- [Background] Chattopadhyay M, Valentine JS. Aggregation of copper-zinc superoxide dismutase in familial and sporadic ALS. Antioxid Redox Signal. 2009 Jul;11(7):1603-14. doi: 10.1089/ars.2009.2536. PMID 19271992
- [Background] Shahrizaila N, Sobue G, Kuwabara S, Kim SH, Birks C, Fan DS, Bae JS, Hu CJ, Gourie-Devi M, Noto Y, Shibuya K, Goh KJ, Kaji R, Tsai CP, Cui L, Talman P, Henderson RD, Vucic S, Kiernan MC. Amyotrophic lateral sclerosis and motor neuron syndromes in Asia. J Neurol Neurosurg Psychiatry. 2016 Aug;87(8):821-30. doi: 10.1136/jnnp-2015-312751. Epub 2016 Apr 19. PMID 27093948
- [Background] Brown RH, Al-Chalabi A. Amyotrophic Lateral Sclerosis. N Engl J Med. 2017 Jul 13;377(2):162-172. doi: 10.1056/NEJMra1603471. No abstract available. PMID 28700839